CLINICAL TRIAL: NCT03501706
Title: Remediation of Elevated Delay Discounting in Mid-life Individuals: A Stage-II Trial
Brief Title: An Assessment of Cognitive Improvement Training Among Mid-life Individuals
Acronym: RehabEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: University of Maryland, Baltimore (Other); University of Florida (Other); Michigan State University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00143274; 7R01AG048904 (NIH)
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Delay Discounting
Keywords: intertemporal tradeoffs; delayed gratification; executive functioning; delay discounting; working memory

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Training (AT) Group (Experimental): Participants will complete four computerized training programs to improve executive function (EF), including Sequenced Recall of Digits - Auditory, Sequenced Reverse Recall of Digits - Auditory, Sequenced Recall of Words - Visual, Verbal Memory - Visual.
  Interventions: Behavioral: Sequenced Recall of Digits--Auditory; Behavioral: Sequenced Reverse Recall of Digits--Auditory; Behavioral: Sequenced Recall of Words--Visual; Behavioral: Verbal Memory--Visual
- Control Training (CT) Group (No Intervention): Participants will complete the four computerized programs relating to executive function (EF), but will be provided with the answer (i.e., without memory requirements). That is, participants in the control condition will not be asked to engage their cognitive functions.

INTERVENTIONS:
Behavioral: Sequenced Recall of Digits--Auditory — Auditory digit sequence AT memory component.
  Arms: Active Training (AT) Group
Behavioral: Sequenced Reverse Recall of Digits--Auditory — Reversed auditory digit sequence AT memory component.
  Arms: Active Training (AT) Group
Behavioral: Sequenced Recall of Words--Visual — Visual word sequence AT memory component
  Arms: Active Training (AT) Group
Behavioral: Verbal Memory--Visual — word recognition AT memory component
  Arms: Active Training (AT) Group

SUMMARY:
Many health-relevant decisions involve intertemporal (now vs. later) tradeoffs. Extensive literature indicates that many negative health and financial consequences suffered in mid-life are linked to adversity and disadvantage during early developmental periods of life. Individuals who continue to engage in these types of unhealthy behaviors despite awareness of the health consequences are exhibiting an inability to delay gratification.

Delay discounting (DD) is quantified in human studies by determining the rate at which an individual discounts a delayed reward, while executive function (EF) is defined as the set of cognitive processes that are responsible for helping individuals manage life tasks and achieve goals. This research will attempt to reduce DD via EF training in a population of mid-life individuals with risk factors established during early-life disadvantage.

DETAILED DESCRIPTION:
Many health-relevant decisions involve intertemporal (now vs. later) tradeoffs, where unhealthy choices involve immediate benefits and delayed costs, compared to healthy choices with immediate costs and delayed benefits. Reinforcement for unhealthy behaviors are immediate, while the reinforcement for healthier alternatives are delayed. Thus individuals who continue to engage in these types of unhealthy behaviors despite awareness of the health consequences are exhibiting an inability to delay gratification.

Delay discounting (DD) is quantified in human studies by determining the rate at which an individual discounts a delayed reward, typically assessed by having subjects choose between a rewards available immediately and a larger reward available following a delay. For the purpose of this study, the investigators define executive function (EF) as the set of cognitive processes that are responsible for helping individuals manage life tasks and achieve goals (e.g., planning, working memory).

The approach of targeting preference for immediate rewards (exhibited by elevated DD) is highly innovative. Multiple studies provide compelling evidence that strengthening EF may decrease DD. Extensive literature indicates that many negative health and financial consequences suffered in mid-life are linked to adversity and disadvantage during early developmental periods of life. By targeting a mechanism of various negative aging-related outcomes (elevated DD), the proposed research may have the novel impact on broadly remediating the health and wellness of mid-life individuals at increased risk for poor consequences due to early-life disadvantage.

This research will attempt to reduce Delay Discounting via Executive Functioning training in a population of mid-life individuals with risk factors established during early-life disadvantage. DD, EF, and associated health behaviors/outcomes will be assessed at baseline, following training, and at 3- and 6-month follow-up. Participants will receive Active EF training, or Control training. Given the established effect of Active training in reducing DD in stimulant-dependent individuals, the study team expect reductions in DD, improvements in EF, and improvements in associated health behaviors/outcomes following Active training and at follow-up, with no improvements in the Control group.

ELIGIBILITY:
Inclusion Criteria:

* Community members in neighborhoods of Baltimore, Maryland
* Participants willing to participate in the 5-7 week program

Exclusion Criteria:

* Participants with a severe substance use disorder according to the DSM-5 with any substance other than tobacco
* Participants with any significant medical or psychiatric condition which the training is not designed for (e.g., traumatic brain injury, dementia, significant learning disability, or schizophrenia)
* Participants with severe depression

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 680 (Estimated)
Dates: Start 2014-11-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Delay Discounting (DD) | Baseline; Week 6-8; Month 3; Month 6
  A binary choice procedure will be conducted on a personal computer to assess relative preference for immediate versus delayed rewards.

SECONDARY OUTCOMES:
Change in Letter Numbering Sequencing (LTC) | Baseline; Week 6-8; Month 3; Month 6
  The participant is given a mixed string of letters and numbers that must then be put into a sequential order of numbers followed by a sequential order of letters.
Change in Hopkins Verbal Learning Test | Baseline; Week 6-8; Month 3; Month 6
  Participants memorize a list of words presented auditorily, then are asked to recall or recognize as many words as possible, either immediately or following a delay.
Change in Tower of Hanoi (ToH) | Baseline; Week 6-8; Month 3; Month 6
  Participants must move the stack of disks from one peg to another while following specific rules.
Change in Iowa Gambling Task | Baseline; Week 6-8; Month 3; Month 6
  Participants are asked to choose to flip cards from one of 4 decks, where each deck is associated with a specific probability of winning and losing some money.

OTHER OUTCOMES:
Change in Timeline Follow-Back | Baseline; Week 6-8; Month 3; Month 6
  Assess relevant point prevalence of alcohol/tobacco/drug use.
Change in The Multidimensional Health Locus of Control | Baseline; Week 6-8; Month 3; Month 6
  An 18-item questionnaire assessing the perception of the underlying causes of health outcomes events.
Change in Chernyshenko Conscientiousness Scale (CCS) | Baseline; Week 6-8; Month 3; Month 6
  CCS is used to assess six facets of conscientiousness, ranking them on a scale of 1-4 with 4 being strongly agree.
Resource Utilization Measure | Baseline; Week 6-8; Month 3; Month 6
  Addresses if individuals accessed healthcare providers in the past thirty days, including visits to doctor's offices or seeing a mental health professional
Change in Patient Activation Measure | Baseline; Week 6-8; Month 3; Month 6
  Assesses how knowledgeable participants are about their health and how they can control it.
Starting the Conversation: Diet Questionnaire | Baseline; Week 6-8; Month 3; Month 6
  Assesses participants' diet
Change in blood pressure | Baseline; Week 6-8; Month 3; Month 6
  systolic and dystolic blood pressure
Change in lipid profile | Baseline; Week 6-8; Month 3; Month 6
  assessing abnormalties in lipids
Change in body mass index | Baseline; Week 6-8; Month 3; Month 6
  body mass index, a ratio of weight (kg) and height (m) will be calculated as kg/m^2
Change in body expired carbon monoxide | Baseline; Week 6-8; Month 3; Month 6
  expired carbon monoxide (parts per million), a measure of recent cigarette smoking
Change in physical activity | Baseline; Week 6-8; Month 3; Month 6
  International Physical Activity Questionnaire (IPAQ) self-reported physical activity assessment

CONTACTS AND LOCATIONS:
Overall Officials: Richard Yi, PhD, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas-Lawrence, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share all de-identified data.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year following publication of the primary outcomes.
Access Criteria: Inquiry with PI

REFERENCES:
- [Derived] Collado A, Felton J, Grunevski S, Doran K, Yi R. Working Memory Training Reduces Cigarette Smoking Among Low-Income Individuals With Elevated Delay Discounting. Nicotine Tob Res. 2022 Apr 28;24(6):890-896. doi: 10.1093/ntr/ntac005. PMID 35018452
- [Derived] Doran K, Collado A, Taylor H, Felton JW, Tormohlen KN, Yi R. Methods to Optimize Recruitment, Participation, and Retention Among Vulnerable Individuals Participating in a Longitudinal Clinical Trial. Res Theory Nurs Pract. 2021 Feb 1;35(1):24-49. doi: 10.1891/RTNP-D-19-00039. PMID 33632921
- [Derived] Felton JW, Collado A, Ingram KM, Doran K, Yi R. Improvement of Working Memory is a Mechanism for Reductions in Delay Discounting Among Mid-Age Individuals in an Urban Medically Underserved Area. Ann Behav Med. 2019 Oct 7;53(11):988-998. doi: 10.1093/abm/kaz010. PMID 30955043